CLINICAL TRIAL: NCT06800625
Title: Manual Versus Sonic-powered Toothbrushing for Plaque Reduction in Patients with Peri-implant Mucositis: Randomized Controlled Trial.
Brief Title: Manual Versus Sonic-powered Toothbrushing for Plaque Reduction in Patients with Peri-implant Mucositis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Niğde Ömer Halisdemir University (Unknown)
Responsible Party: Principal Investigator, Selcen Ozcan Bulut, asist. prof, Hacettepe University
Other Study IDs: 2023/15
Record Dates: First submitted 2025-01-22; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Toothbrushing; Periimplant Diseases
Keywords: Biofilm; Dental İmplant; Peri-implant mucositis; Toothbrushing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1.gruop: Manuel toothbrusing: Patients with peri-implant mucositis were instructed to use manuel toothbrushing for plaque reduction.
- 2. group: sonic-powered toothbrushing: Patients with peri-implant mucositis were instructed to use sonic-powered toothbrushing for plaque reduction.

SUMMARY:
Aim: To compare the effect of manual and sonic-powered toothbrushing on biofilm control in patients with peri-implant mucositis.

Materials and methods: The study was completed with a total of 41 patients, 21 in the sonic tooth brushing group and 20 in the manual tooth brushing group. The patients' baseline, 3rd-month, 6th-month and 9th-month periodontal examination data (Modified Gingival İndex (MGI), Modified plaque index (MPI), Bleeding on the probing index (BOP), Pocket depth (PD), Gingival Recession (GR) and Gingival Biotype (GB)) were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Bleeding on probing around the implant
2. No bone loss around the implant in the radiograph
3. Having adequate keratinized gingiva around the implant
4. The presence of an implant prosthesis that was installed at least three months previously
5. No systemic disease
6. no smoke
7. No use of antibiotic medications within the previous three months

Exclusion Criteria:

1. Patients with missing data and who do not allow data use
2. Smoker
3. Data from pregnant and lactating patients
4. Pocket depth around the implant is ≥ 5
5. Patients with peri-implantitis (bone loss around the implant)
6. Patients with insufficient attached gingiva around the implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to Niğde Ömer Halisdemir University Faculty of Dentistry Periodontics Clinic between 15.04.2023 and 15.06.2023 for the control of dental implants and/or periodontal treatment, volunteered to participate in the study and met the following criteria were included in the study. Written consent was obtained from volunteer patients for the research.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Modified Gingival İndex (MGI) | baseline, 3rd-month, 6th-month and 9th-month
  In order to determine the degree of inflammation in the surrounding soft tissue of the implants, mGI score is obtained from four regions: mesial, distal, buccal and palatal. The mGI score for each implant is determined by adding the values and dividing by 4.
  Scoring is done as follows; 0: No bleeding when probing around the implant with a periodontal probe l: There is a point isolated bleeding on probing. 2: On probing, there is bleeding forming a red line along the mucosal margin. 3: There is intense bleeding on probing.
Modified plaque index (MPI) | baseline, 3rd-month, 6th-month and 9th-month
  This index, which is used to determine the surface cleanliness of implants, is measured from 4 regions of the implants: mesial, distal, buccal and palatal, taking into account the following criteria. The mPI score for each implant is determined by adding the obtained values and dividing by 4.
  Scoring is done as follows; 0: No record. l: Presence of plaque in the implant sulcus that can be detected with the probe tip. If there is a roughened implant surface in this area, at least "1" value is given.
  2: Presence of visible plaque. 3: Presence of soft attachment on the implant surface c. Bleeding on Probing Index (BOP) Approximately 20 seconds after moving the periodontal probe inside the periodontal pocket, it is evaluated whether there is bleeding. If there is bleeding, the score of that area is recorded as (+), otherwise it is recorded as (-).

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Dentistry Faculty, Periodontology Department, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided